CLINICAL TRIAL: NCT02285894
Title: Can 10 Seconds Inspiratory Hold Open Atelectasis in Mechanically Ventilated Patients? A Pilot Study.
Brief Title: Can 10 Seconds Inspiratory Hold Open Atelectasis in Mechanically Ventilated Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/375 (REK)
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inspiratory hold (Experimental): Mechanical inspiratory pressure held for 10 seconds at a time.
  Interventions: Other: Inspiratory hold

INTERVENTIONS:
Other: Inspiratory hold — Sustainment of the ventilators inspiratory pressure for 10 seconds at a time

SUMMARY:
This study evaluates whether sustaining inspiratory pressure for 10 seconds at a time can open collapsed lung areas in non-dependant regions of the lung in mechanically ventilated patients.

DETAILED DESCRIPTION:
Collapse of lung volume, atelectasis, is a common complication in sedated and mechanically ventilated patients. In adults the atelectasis occur mainly in the dependant areas of the lung. In this study the investigators examine whether these atelectasis can be opened by repeatedly sustaining the inspiratory pressure for 10 seconds when the patient has been positioned so that the atelectasis is located in a non-dependant position. Furthermore, the investigators examine how many times the inspiratory pressure needs to be sustained before the atelectasis is opened and at what pressure.

ELIGIBILITY:
Inclusion Criteria:

* Continuously or intermittently mechanically ventilated with artificial airway (endotracheal tube or tracheostomy tube)
* Pressure controlled or pressure supported ventilator mode
* PEEP ≤ 12 cm H2O, registered peak pressure ≤ 32 cm H2O
* Non-ventilated lung regions according to E.I.T. measurements
* Richmond Agitation Score 0 -(-5)
* Circulatory stable or stabilized

Exclusion Criteria:

* Pregnancy
* BMI > 50
* Pacemaker or other electrically active implants
* Skin lesions, wounds or bandages on chest area where E.I.T. belt needs to be placed
* Undrained pneumothorax
* Pulsating air-mattress
* Unstable skeletal injury to spinal column
* Recent brain injury or spinal chord injury
* Recent injury to heart, to major blood vessels in chest, to major airways or to the oesophagus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Ventilation in previously non-ventilated lung tissue | During intervention and for 30 minutes after ended intervention
  Registered using electrical impedance tomography, E.I.T., via PulmoVista500 by Dräger Medical

CONTACTS AND LOCATIONS:
Overall Officials: Nina K Vøllestad, Dr.Scient, Principal Investigator — University of Oslo; Harald Noddeland, PhD, MD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo university Hospital, Ullevål, Oslo, Oslo County, Norway